CLINICAL TRIAL: NCT05708677
Title: A Long-Term Extension Study for Participants Previously Treated With EB-101 for the Treatment of Recessive Dystrophic Epidermolysis Bullosa (RDEB)
Brief Title: A Long-Term Extension Study for Participants Previously Treated With EB-101 for the Treatment of RDEB
Status: Enrolling by invitation | Type: Observational
Sponsor: Abeona Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: EB-101-LT-001
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: RDEB

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Long-Term Extension: This study will follow one group of participants who were enrolled in a previous EB-101 study.
  Interventions: Biological: EB-101

INTERVENTIONS:
Biological: EB-101 — This is non-interventional and follows patients treated with EB-101
  Other Names: pz-cel

SUMMARY:
A Long-Term Extension Study for Participants Previously Treated with EB-101 for the Treatment of Recessive Dystrophic Epidermolysis Bullosa (RDEB)

DETAILED DESCRIPTION:
This is an open-label, long-term, follow-up study in participants from prior interventional trials involving surgical application of gene-corrected keratinocyte sheets (EB-101) for the treatment of RDEB wound sites. Up to 22 participants will be enrolled in this study, with follow-up through at least 5 years post treatment. Patient-reported outcomes and safety will be assessed throughout the study, and where applicable, compared to Baseline of the preceding interventional EB-101 trial. Upon completion, participants will transfer to an annual monitoring program for additional 10 years of phone visits.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give consent/assent;
* If under the age of 18, guardian(s) is/are willing and able to give consent;
* Prior study treatment with EB-101.

Exclusion Criteria:

* Inability to properly follow protocol as determined by the Principal Investigator

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with previous EB-101 treatment
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2021-02-09 (Actual); Primary Completion 2036-02 (Estimated); Study Completion 2036-08 (Estimated)

PRIMARY OUTCOMES:
Wound Closure | 5 years
  Proportion of RDEB wounds with healing ≥50%, ≥75%, and 100% at all clinic visits up to Month 54 as determined by direct investigator assessment.
Pain Reduction | 5 years
  Pain reduction assessed by Wong-Baker FACES scale at all clinic visits up to Month 54.
Itch Severity | 5 years
  Longitudinal change of Itch severity scores assessed at all clinic visits up to Week 54.
Zarit Burden Interview | 5 years
  Longitudinal change of Zarit Burden Interview Short Form (ZBI-12) for caregiver scores related to wound care, assessed at all clinic visits up to Month 54.
Quality of Life | 5 years
  Quality of Life in Epidermolysis Bullosa (QOLEB) scores assessed at all clinic visits up to Month 54.
Caregiver Global impression of Pain | 5 years
  Caregiver Global impression of Pain (CrGI-Pain) scores assessed at all clinic visits up to Month 54.
Wound Infection and Adverse Events | 5 years
  The number of participants and wounds that have an infection or any related adverse event.
The number of treatment-emergent adverse events. | 5 years
  The number of treatment-emergent adverse events.
Serious Adverse Events | 5 years
  The number of participants and wounds that result in hospitalization (serious adverse event [SAE]).
Incidence of squamous cell carcinoma. | 5 years
  Incidence of squamous cell carcinoma.
Replication-competent retrovirus (RCR) status | 5 years
  Replication-competent retrovirus (RCR) status

CONTACTS AND LOCATIONS:
Overall Officials: Angela Iheanacho, MS, Study Director — Abeona Therapeutics, Inc; Sarah Abdelwahab, MD, Study Director — Abeona Therapeutics, Inc
Locations (2):
- United States (2):
  - Stanford University, Redwood City, California
  - University of Massachusetts Medical School, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided